CLINICAL TRIAL: NCT02360384
Title: A Randomised Controlled Trial to Validate the Use of Caecal pH Measurement as a Biomarker in Irritable Bowel Syndrome
Brief Title: Caecal pH as a Biomarker for Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Wingate Institute of Neurogastroenterology (Other)
Responsible Party: Principal Investigator, Adam Farmer, Consultant gastroenterologist, Wingate Institute of Neurogastroenterology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: WMC1
Record Dates: First submitted 2015-01-25; First posted 2015-02-10 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: wireless motility capsule
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — linaclotide; FODMAP Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sham diet (Placebo Comparator): The placebo intervention will be healthy eating advice in patients with irritable bowel syndrome of the alternating subtype for 28 days.
  Interventions: Drug: Linaclotide
- Lincalotide (Active Comparator): All patients with constipation predominant IBS will receive linaclotide 280mcg po od for 28 days.
  Interventions: Drug: Linaclotide
- FODMAP diet (Experimental): The FODMAP diet will be introduced in patients with irritable bowel syndrome of the alternating subtype for 28 days.
  Interventions: Dietary Supplement: FODMAP diet

INTERVENTIONS:
Drug: Linaclotide — Linaclotide 290mcg po od in all patients with irritable bowel syndrome with constipation.
  Other Names: Constella
  Arms: Lincalotide; Sham diet
Dietary Supplement: FODMAP diet — Patients with irritable bowel syndrome with alternating bowel habit will be commenced on the either the low FODMAP diet or a control healthy eating diet.
  Arms: FODMAP diet

SUMMARY:
Irritable bowel syndrome is common. Currently, it is a diagnosis of exclusion. There is increasing evidence of the importance of the microbiota in the pathophysiology of this disorder. However, it has been challenging to measure the "activity" of the microbiota in vivo as much of the GI tract is inaccessible. Fermentation by the microbiota occurs in the colon, a by product of which are short chain fatty acids. Measuring pH in the colon could potentially act as a surrogate marker of fermentation. The investigators are undertaking a randomised controlled trial in patients with IBS measuring the pH in the digestive tract using a wireless motility capsule at baseline and in response to dietary changes in patients with diarrhoea predominant IBS and in response to linaclotide in those with constipation predominant IBS to ascertain the effect of these interventions on the microbiota and clinical outcomes.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is an extremely common condition. Between 1.9 and 3.6 million patients consult a healthcare professional for IBS each year in the UK (1). The total population prevalence is much higher as most IBS sufferers are non-consulters due to the perceived lack of effective treatments. IBS can be sub-classified based upon predominating bowel habit, i.e. constipation predominant (IBS-C), alternating bowel habit (IBS-A) or diarrhoea predominant (2). In recent years, several efficacious treatment approaches have been applied to IBS including dietary interventions (low fibre and low fermentable oligosaccharides, disaccha¬rides, monosaccharides and polyols (FODMAP)), probiotics (VSL#3) and pharmacological agents (linaclotide) (3). Whilst each of these treatment approaches have shown efficacy, it is clear that further refinement of the IBS diagnostic algorithm is required to better target therapies in order to overcome the inherent heterogeneity within the IBS population.

Bloating and distension are both common and vexatious symptoms in a proportion of IBS patients. Bloating is largely regarded as a subjective sensation of abdominal swelling, whereas distension refers to an observable increase in abdominal girth. Bloating is associated with a reduction in quality of life, is a cause for healthcare seeking and represents a considerable challenge to manage effectively.

The anaerobic breakdown of carbohydrates and protein by bacteria, largely occurring within the proximal colon, is through a process known as fermentation, the principal products of which are short chain fatty acids (SCFA). One of the proposed mechanisms of bloating and distension is colonic dysbiosis and subsequent mal-fermentation. This has been supported by data which show that a large proportion of IBS patients improve symptomatically when restricting their diet to an 'elemental' formula for 2-4 weeks thus reducing the amount of fermentable material in the intestinal lumen.

The direct in vivo measurement of SCFA concentrations in the human proximal colon is technically difficult and invasive. Given that the degree of bacterial fermentation is directly proportional to the concentration of SCFA, the measurement of segmental intra-colonic pH is an inverse surrogate proxy of the degree of fermentation occurring within that territory. We have recently shown that measurement of caecal pH using the wireless motility capsule (WMC) in IBS and control patients is both technical feasible and able to differentiate between the two populations (4).

Our study showed that caecal pH is significantly lower in IBS when compared to controls thus supporting the concept that mal-fermentation is contributing to IBS symptomatology. Importantly, we have also shown that caecal pH is correlated with inhibition of caecal contractility which has led us to propose the idea that 'caecoparesis' maybe the long sought after alteration in motor function which differentiates IBS patients from healthy participants and explains why IBS preferentially experience pain in the right colon and upper abdomen in response to balloon distension.

TRIAL OBJECTIVES The primary aim of this study is to demonstrate that caecal pH is a sensitive and reliable biomarker of caecal fermentation in IBS and that normalisation of the caecal pH environment will correlate with symptomatic improvement in IBS patients. We hypothesise that normalisation of the caecal pH environment with either dietary intervention or linaclotide will correlate with symptomatic improvement in IBS patients. To achieve this we will recruit a cohort of Rome III defined IBS patients and sub-divide them into the appropriate IBS type based on symptoms. We will then characterise their phenotype in terms of gastro-intestinal physiology (WMC + lactulose hydrogen breath test) and psychological profile. They will then be allocated to one of (2 or 3) treatment arms (control diet, low FODMAP diet, control diet + linaclotide). Each treatment arm will last for 28 days after which WMC will be repeated and symptoms assessed. Secondary aims will include characterising motility and transit in IBS-sub groups, determining the effect of the interventions of motility and transit, comparison of ileal and caecal pH profiles with hydrogen / methane breath testing data and comparison of symptom change and physiological assessment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide Informed written consent
* Age (18-65 years old)
* Male and female patients with irritable bowel syndrome of the alternating or constipation subtype.

Exclusion Criteria:

* Any inclusion criteria not met
* Participants unable to provide informed consent.
* Participants on any medications that may influence gastrointestinal motility (e.g. beta-agonists).
* Pregnancy.
* Recent antibiotic use in the preceding 4 weeks.
* Recent probiotic use in the last 2 weeks, concurrent use of promotile medications.
* Participants with IBS-C who are already taking linaclotide or have known hypersensitivity to linaclotide.
* History of a systemic disorder with known gastrointestinal manifestations (such as diabetes mellitus, connective tissue disorders etc.) and previous gastrointestinal tract surgery will be treated as criteria for exclusion. Specific contraindications to WMC are dysphagia, recent abdominal surgery, Crohn's disease, planned MRI and diverticulitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the change in pH around the ileocaecal valve in response to dietary intervention or linaclotide. | 28 days
  Change in pH around the ileocaecal valve using the wireless motility capsule in response to the dietary intervention and linaclotide

SECONDARY OUTCOMES:
Change in caecal pH and its association with the degree in symptomatic improvement using the IBS-symptom scale | 28 days
  The change in caecal pH association and it is association with the magnitude of improvement in symptoms using the validated IBS-SSS questionnaire
Motility patterns and transit in subtype IBS patients, according to the Rome III criteria, using the wireless motility capsule | 1-2 days
The effect of the interventions on symptoms using the validated questionnaires of IBS-SSS | 28 days
The effect of the interventions on quality of life measures using the validated Eq-5D | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Adam D Farmer, PhD MRCP, Principal Investigator — Wingate Institute of Neurogastroenterology
Locations (1):
- Wingate Institute of Neurogastroenterology, London, London, United Kingdom

REFERENCES:
- [Background] Farmer AD, Mohammed SD, Dukes GE, Scott SM, Hobson AR. Caecal pH is a biomarker of excessive colonic fermentation. World J Gastroenterol. 2014 May 7;20(17):5000-7. doi: 10.3748/wjg.v20.i17.5000. PMID 24803812